CLINICAL TRIAL: NCT06134414
Title: A Multi-center, Randomized, Parallel, Open-label Clinical Phase II Study, to Evaluate the Efficacy and Safety of MY008211A in Adult Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients With Signs of Active Hemolysis
Brief Title: Study of Safety and Efficacy of MY008211A in in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MY008211A-PNH-2-01-F
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 MY008211A low dose (Experimental): Participants will receive MY008211A at a dose of 400 mg orally b.i.d
  Interventions: Drug: MY008211A tablets
- Arm 2 MY008211A high dose (Experimental): Participants will receive MY008211A at a dose of 600 mg orally b.i.d
  Interventions: Drug: MY008211A tablets

INTERVENTIONS:
Drug: MY008211A tablets — dose 1 (400 mg BID) and dose 2 (600 mg BID) in a 1:1 ratio by central randomization
  Other Names: MY008211A

SUMMARY:
The main purpose of this study is to evaluate the efficacy of MY008211A in adult patients with PNH, showing signs of active hemolysis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether MY008211A is efficacious and safe for the treatment of PNH patients who are naïve to complement inhibitor therapy, including anti-C5 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age and BMI ≥ 18.0 kg/m2 with a diagnosis of PNH confirmed by high-sensitivity flow cytometry with clone size ≥ 10%.
* Mean hemoglobin level <100 g/L.
* LDH > 1.5 x Upper Limit of Normal (ULN).
* Vaccination against Neisseria meningitidis infection is required prior to the start of study treatment. If not received previously, vaccination against Streptococcus pneumoniae and Haemophilus influenzae infections should be given.

Exclusion Criteria:

* Patients with reticulocytes <100x10^9/L; platelets <30x10^9/L; neutrophils <0.5x10^9/L.
* Were using a complement inhibitor before the first administration of MY008211A tablets or had discontinued a previous complement inhibitor for less than five half-lives or 120 days, whichever was the longest.
* History of recurrent invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus.
* Known or suspected hereditary complement deficiency.
* Previous bone marrow or hematopoietic stem cell transplantation.
* Previous splenectomy.
* A history of malignancy within 5 years before screening, except cured local basal cell carcinoma of the skin and carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with an increase in hemoglobin concentration ≥ 20 g/L from baseline among subjects who do not receive RBC transfusion after 4 weeks of dosing | Day 70
  Proportion of participants achieving a sustained increase from baseline in hemoglobin levels of ≥ 20 g/L assessed , in the absence of red blood cell transfusions

SECONDARY OUTCOMES:
The proportion of patients with an increase in hemoglobin ≥ 20 g/L from baseline among those without RBC transfusion | Day14, 21, 28, 42, 56
  The proportion of patients with an increase in hemoglobin ≥ 20 g/L from baseline among those without RBC transfusion
The proportion of patients with hemoglobin ≥ 120 g/L among those without RBC transfusion | Day14, 21, 28, 42, 56 and 70
  The proportion of patients with hemoglobin ≥ 120 g/L among those without RBC transfusion
Change in hemoglobin concentration from baseline in patients without RBC transfusion | Day14, 21, 28, 42, 56 and 70
  Change in hemoglobin concentration from baseline in patients without RBC transfusion
Change in LDH level from baseline | Day7, 14, 21, 28, 42, 56 and 70
  Change in LDH level from baseline
The proportion of patients with hemolysis controlled | Day7, 14, 21, 28, 42, 56 and 70
  The proportion of patients with hemolysis controlled (defined as LDH < 1.5 ULN)
Change in reticulocyte count from baseline in patients without RBC transfusion | Day7, 14, 21, 28, 42, 56 and 70
  Change in reticulocyte count from baseline in patients without RBC transfusion
Change in indirect bilirubin level from baseline | Day7, 14, 21, 28, 42, 56 and 70
  Change in indirect bilirubin level from baseline
The proportion of patients without RBC transfusion | Day14, 21, 28, 42, 56 and 70
  The proportion of patients without RBC transfusion
Change in the average weekly amount of RBC transfused during the efficacy observation period | Day70
  Change in the average weekly amount of RBC transfused during the efficacy observation period compared with that pre-dose
Change From Baseline in FACIT-Fatigue Questionnaire | Day7, 14, 21, 28, 42, 56 and 70
  Change from baseline in FACIT-Fatigue scores. The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
Changes from baseline in alternative complement pathway activity | Day14, 28, 56 and 70
  Alternative complement pathway activity measured by the WIESLAB® kit.
Change in the amount of fragment Bb of CFB in plasma from baseline | Day14, 28, 56 and 70
  Bb fragment cleaved by factor B of complement.
Change in the level of PNH RBC clones from baseline in patients without RBC transfusion. | Day70
  Change from baseline in the level of PNH red cell clones.
Incidence of Adverse Events (AEs) between Day 1 and Day 70 | Day 70
  Adverse Events (AEs)